CLINICAL TRIAL: NCT04993430
Title: A Phase 1, Single Arm, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability and Pharmacokinetic of HRS8807 Monotherapy and in Combination With SHR6390 in Subjects With ER-Positive, HER2-Negative Metastatic or Locally Advanced Breast Cancer
Brief Title: A Phase 1 Study of HRS8807 Monotherapy and in Combination With SHR6390 in Subjects With ER-Positive, HER2-Negative Metastatic or Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS8807-I-101
Record Dates: First submitted 2021-07-20; First posted 2021-08-06 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: ER-Positive, HER2-Negative Breast Cancer

STUDY DESIGN:
Intervention Model Description: HRS8807 monotherapy and in combination with SHR6390
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): HRS8807 monotherapy dose escalation
  Interventions: Drug: HRS8807
- Group B (Experimental): HRS8807 monotherapy dose expansion
  Interventions: Drug: HRS8807
- Group C (Experimental): HRS8807 in combination with SHR6390 dose escalation
  Interventions: Device: HRS8807、SHR6390
- Group D (Experimental): HRS8807 in combination with SHR6390 dose expansion
  Interventions: Drug: HRS8807、SHR6390

INTERVENTIONS:
Drug: HRS8807 — HRS8807 monotherapy
  Arms: Group A
Drug: HRS8807 — HRS8807 monotherapy
  Arms: Group B
Device: HRS8807、SHR6390 — HRS8807 in combination with SHR6390
  Arms: Group C
Drug: HRS8807、SHR6390 — HRS8807 in combination with SHR6390
  Arms: Group D

SUMMARY:
The study is to assess safety and tolerability of HRS8807 monotherapy and in combination with SHR6390 in subjects with metastatic or locally advanced breast cancer in order to estimate the Dose-Limiting Toxicity (DLT), Maximum Tolerated Dose (MTD) and select the Recommended Phase 2 Dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of metastatic or locally advanced breast cancer; Histologically proven diagnosis of ER-positive, HER2-negative;
2. At least 1 line of endocrine therapy in the metastatic or advanced setting that had progressed or intolerance; ≤ 2 lines of chemotherapy for metastatic or advanced disease;
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1;
4. Expected survival of more than 3 months.

Exclusion Criteria:

1. All patients in monotherapy and or in combination wih phase who are known allergic to HRS8807 or SHR6390 ingredient;
2. Presence of symptomatic metastatic visceral disease ;
3. Patients with known active brain metastases;
4. Clinically serious cardiovascular disease;
5. Abnormal electrocardiographic (ECG) with clinical significancy by investigator judgement;
6. Abnormal thyroid function laboratory results;
7. Active infection or unexplained fever >38.5℃ during screening period or on the day of the first dose.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD | Change From Baseline at 28 days
  Maximum Tolerated Dose (MTD) of HRS8807 monotherapy and in combination with SHR6390
RP2D | Change From Baseline at 28 days
  select the Recommended Phase 2 Dose (RP2D) of HRS8807 monotherapy and in combination with SHR6390
Adverse events (AE) and serious AE (SAE) | Up to 30 days after end of treatment
  AEs and SAEs as characterized by frequency and severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE version 5.0]).

SECONDARY OUTCOMES:
Tmax of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
Cmax of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
AUC0-t of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
AUC0-∞ of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
t1/2 of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
Vz/F of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
CL/F of HRS8807 and the major metabolite after single dose of HRS8807 | Day 1, Day 2, Day 3 of single dose (3 days before Cycle1)
Tmax,ss of HRS8807 and the major metabolite after multiple dose administration of HRS8807 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Cmax,ss of HRS8807 and the major metabolite after multiple dose administration of HRS8807 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Cmin,ss of HRS8807 and the major metabolite after multiple dose administration of HRS8807 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Rac of HRS8807 and the major metabolite after multiple dose administration of HRS8807 | Cycle 1 Day 14, Day 15, each cycle is 28 days
AUCss of HRS8807 and the major metabolite after multiple dose administration of HRS8807 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Tmax of HRS8807, the major metabolite and SHR6390 after single dose administration of HRS8807 and SHR6390 | Cycle 1 Day 1, Day 2, each cycle is 28 days
Cmax of HRS8807, the major metabolite and SHR6390 after single dose administration of HRS8807 and SHR6390 | Cycle 1 Day 1, Day 2, each cycle is 28 days
AUC0-t of HRS8807, the major metabolite and SHR6390 after single dose administration of HRS8807 and SHR6390 | Cycle 1 Day 1, Day 2, each cycle is 28 days
Tmax,ss of HRS8807, the major metabolite and SHR6390 after multiple dose administration of HRS8807 and SHR6390 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Cmax,ss of HRS8807, the major metabolite and SHR6390 after multiple dose administration of HRS8807 and SHR6390 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Cmin,ss of HRS8807, the major metabolite and SHR6390 after multiple dose administration of HRS8807 and SHR6390 | Cycle 1 Day 14, Day 15, each cycle is 28 days
AUCss of HRS8807, the major metabolite and SHR6390 after multiple dose administration of HRS8807 and SHR6390 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Rac of HRS8807, the major metabolite and SHR6390 after multiple dose administration of HRS8807 and SHR6390 | Cycle 1 Day 14, Day 15, each cycle is 28 days
Objective Response Rate (ORR) | baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered participant
Duration of Response (DoR) | baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered participant
Progression Free Survival (PFS) | baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered participant

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided